CLINICAL TRIAL: NCT01455025
Title: A Phase 1, Dose Escalation Study of Plerixafor in Combination With Induction and Consolidation Chemotherapy in Patients With Relapsed Acute Myeloid Leukemia
Brief Title: Study in Plerixafor and Granulocyte-colony Stimulating Factor Patients With Relapse Acute Myeloid Leukemia
Acronym: PRIMAL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no recruitment on time
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Primal study
Record Dates: First submitted 2011-06-24; First posted 2011-10-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Plerixafor granulocyte-colony stimulating factor; Chemotherapy in relapse; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plerixafor granulocyte-colony stimulating factor (Experimental): 4 steps of plerixafor doses from 240 to 480 microgram/kg per day concomitant with GCSF and chemotherapy 3 to 6 evaluable patients will be enrolled at each dose level in a modified 3 + 3 design.
  Interventions: Drug: Plerixafor granulocyte-colony stimulating factor

INTERVENTIONS:
Drug: Plerixafor granulocyte-colony stimulating factor — Induction phase Plerixafor IV from D1 to D3 and from D8 to D10, granulocyte-colony stimulating factor IV 5 μg/kg/day from D1 to D10, Intravenous daunorubicin 60 mg/m2/day from D1 to D3 Cytarabine 500 mg/m2/day continuous infusion over 24h from D1 to D3 followed by cytarabine 2-hour bolus of 1000 mg/m2/12h from D8 to D10.
  Consolidation phase Plerixafor at D1, D3 and D5, granulocyte-colony stimulating factor IV 5 μg/kg/day from D1 to D5, Cytarabine continuous infusion of 3-h bolus of 3000 mg/m2/12h D1, D3 and D5
  Other Names: Plerixafor G CSF

SUMMARY:
This is a phase 1, dose escalation study of Plerixafor in combination with granulocyte-colony stimulating factor , Daunorubicin and Cytarabine in adults patients with relapsed acute myeloid leukemia .

DETAILED DESCRIPTION:
The Primary objective is to determine the maximal tolerated dose and Recommended Phase 2 Dose of plerixafor when used in combination with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine during induction therapy Then determine the tolerability of plerixafor administered in combination with G-CSF and cytarabine during consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Myeloid Leukemia in first relapse with first response duration > 9 months.
* Age between 18 and 65 years.
* Treatment with hydroxyurea or purinethol is allowed if discontinued at least 24 hours before the start of study treatment.
* White blood count less than 30 x 109/L
* Left ventricular ejection fraction more than 50% on echocardiography or multigated acquisition scan or similar radionuclide angiographic scan.
* Total bilirubin less than 1.5 x upper limit of normal= ULN or AST and ALT less than 2.5 x ULN or gammaGT less than 2.5 x ULN.
* Serum creatinine less than 1.5 x ULN and/or creatinine clearance more than 50 ml/mn.
* ECOG performance status less than 2
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Absence of pregnancy or lactation
* Affiliated to French social security system or similar
* Signed informed consent

Exclusion Criteria:

* AML evolving from MPD and/or secondary AML
* Patients treated with more than 270 mg/m2 of daunorubicin during first line therapy.
* Have any of the following within the last 9 months :
* Unstable supraventricular arrhythmia or patient with a pace-maker
* Any ventricular arrhythmia
* Congestive heart failure
* Myocardial infarction, ischemia, stable coronary disease or angina pectoris
* Syncope with a known cardiovascular etiology
* Known hypersensitivity or contra-indication to drugs used in the protocol = G-CSF, daunorubicin, cytarabine or to excipients.
* Previous treatment with plerixafor.
* Previous hematopoietic stem cell transplantation = Allologous or autologous.
* White blood count more than 30 x 109/L despite treatment with hydroxyurea or purinethol.
* Treatment with chemotherapy or G-CSF within 3 months of screening.
* Uncontrolled active infection.
* Uncontrolled arrythmia
* Grade more than 3 renal dysfunction with serum creatinine more than 1.5 x ULN and/or creatinine clearance less than 50 ml/mn.
* Significant neurologic grade more than 2 or psychiatric disorder, dementia or seizures.
* Clinical symptoms suggesting active central nervous system leukemia.
* Pre-existing disorder predisposing the patient to serious or life-threatening infections = cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder or cytopenia
* Thrombocytopenia refractory to platelet transfusion
* Anticoagulant therapy
* Severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock or disseminated intravascular coagulation.
* Thrombocytopenia refractory to platelet transfusion.
* Prior total body irradiation more than 10 Gy.
* Known HIV, Hepatitis B or C positivity.
* Participation into a clinical study of an investigational agent within 14 days before study entry.
* Pregnancy or breastfeeding
* Adult patient protected by law
* Concurrent treatment with any other anti-cancer therapy except hydroxyurea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
maximal tolerated dose | 40 days
  4 steps of plerixafor doses from 240 to 480 microgram per kilogram per day concomitant with granulocyte-colony stimulating factor and chemotherapy Three to 6 evaluable patients will be enrolled at each dose level in a modified 3 + 3 design.

SECONDARY OUTCOMES:
safety and tolerability of plerixafor in combination with granulocyte-colony stimulating factor and chemotherapy | 9 months
  Number of Adverse Events and Serious Adverse Events :examined at each dose level by the Independent Data safety Monitoring Board
Efficacy of plerixafor on leukemic blasts | 10 Days
  study of the drop of leukemic blasts blood rate
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 2 months
  -Minimal Residual Disease level after first consolidation
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 5 weeks
  - Time to remission
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 3 months
  -Rate of patients able to proceed to hematopoietic stel cell transplantation
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 9 months
  -disease free survival
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 9 months
  -event free survival
Efficacy of combination plerixafor with granulocyte-colony stimulating factor, Daunorubicin and Cytarabine | 9 months
  overal survival

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD PD, Principal Investigator — ALFA; Didier BOUSCARY, MD PD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Xavier THOMAS, Lyon, France

REFERENCES:
- See also: FILO website — http://www.filo-leucemie.org